CLINICAL TRIAL: NCT02923596
Title: Retrospective Study of Keloid Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tirgan, Michael H., M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: Tirgan 16-01
Record Dates: First submitted 2016-09-12; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Keloid
Keywords: Keloid
MeSH Terms: conditions — Keloid | interventions — Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with Ear Keloids: Records of Patients with Ear Keloids will be reviewed. Data and photographs will be analysed.
  Interventions: Procedure: History of prior Surgery; Radiation: History of Radiation Therapy
- Patients with Neck Keloids: Records of Patients with Neck area Keloids will be reviewed. Data and photographs will be analysed.
  Interventions: Procedure: History of prior Surgery; Radiation: History of Radiation Therapy
- Patients with Scalp Keloids: Records of Patients with Scalp Keloids will be reviewed. Data and photographs will be analysed.
  Interventions: Procedure: History of prior Surgery; Radiation: History of Radiation Therapy

INTERVENTIONS:
Procedure: History of prior Surgery — History of prior Surgery will be reviewed
  Other Names: Surgery
Radiation: History of Radiation Therapy — History of prior radiation therapy will be reviewed
  Other Names: Radiation Therapy

SUMMARY:
Purpose of this retrospective study is to review and analyze the information and data that has been already been generated during the course of routine practice of medicine by the investigators from 2007 up until Sept 1, 2016 from keloid patients who have sought medical care or medical advice for their keloid disorder.

DETAILED DESCRIPTION:
To retrospectively review and analyze clinical data that has already been collected from keloid patients including photographs taken of keloid lesions during routine practice of medicine by the investigators 1) To better understand natural history of keloid disorder (KD), 2)To determine the ethnic incidence and prevalence of keloid, 3) To determine the rate of familial keloids, 4) To determine response to different treatment modalities, 5) To determine risk factors for development and worsening of keloid lesions.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have at least one keloid lesion.
* Availability of photographic documentation of keloid lesion(s).

Exclusion Criteria:

* Lack of photographic documentation of keloid lesion(s)
* Lack of demographic data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a diagnosis of keloid
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-09; Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Rate of development of massive, semi-massive and large Keloids | 1-5 years after surgery
  Keloid Recurrence after surgery is a real-world outcome, one that takes time to develop. Study will intend to explore the long term rate of keloid recurrence after surgery. This rate will be reported as percentage of patients who undergo surgery and end up with developing a massive, semi-massive or large recurrent keloid

SECONDARY OUTCOMES:
Rate of poor aesthetic outcome after ear surgery | 1-5 years after surgery
  Surgical intervention often results in loss of ear tissue and poor aesthetic outcome. Although fully expected, the actual rates of this outcome is unknown. Study intends to report the actual rate of disfigurement and poor aesthetic outcome after ear surgery for removal of keloid lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Tirgan, MD, Study Chair — Keloid Research Foundation
Locations (2):
- United States (2):
  - Michael H. Tirgan MD, New York, New York
  - Texas Institute of Dermatology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes